CLINICAL TRIAL: NCT05212610
Title: Assessing Safety of COVID-19 mRNA Vaccine Administration in the Setting of a Previous Adverse Reaction
Brief Title: Assessing Safety of Coronavirus Infection (COVID-19) Messenger RNA (mRNA) Vaccine Administration in the Setting of a Previous Adverse Reaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Wallace Foundation (Other)
Responsible Party: Principal Investigator, James Baker Jr MD, Professor of Internal Medicine in Allergy/Clinical Immunology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00206480
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Corona Virus Infection
Keywords: mRNA vaccine; Adverse reactions; Vaccine re-challenge; Allergic reactions; Long COVID infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Hypersensitivity | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pfizer-BioNTech mRNA COVID-19 vaccine (Experimental): Subject will receive an initial or additional dose of the Pfizer-BioNTech (Comirnaty) mRNA COVID-19 vaccine
  Interventions: Biological: Pfizer-BioNTech mRNA COVID-19 vaccine

INTERVENTIONS:
Biological: Pfizer-BioNTech mRNA COVID-19 vaccine — Participants will receive an initial or additional dose of a highly protective COVID-19 mRNA vaccine for the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus in an environment where the investigators and staff are experienced in the care of patients with allergic reactions.
  Other Names: Comirnaty

SUMMARY:
This study will evaluate the safety of administering an additional dose of an mRNA COVID-19 vaccine or mRNA bivalent COVID-19 booster vaccine to individuals who have had adverse reactions to a previous dose or administering an initial dose of an mRNA COVID-19 vaccine to individuals with a personal history of allergic reaction. In addition, this study will evaluate the safety of administering an initial or additional dose or bivalent booster of an mRNA COVID-19 vaccine to individuals experiencing an adverse reaction to a natural COVID-19 infection ("long COVID").

Eligible participants enrolled in this trial will receive an initial or additional dose of either the Pfizer-BioNTech COVID-19 bivalent vaccine or the Moderna COVID-19 bivalent vaccine. Participants will also be required to have 1-2 in person visits along with phone call follow up visits.

We hypothesize that individuals who have had adverse reactions to a previous dose of an mRNA COVID-19 vaccine will tolerate an additional dose of the primary mRNA vaccine or bivalent booster, as indicated, and those with a personal history of allergic reaction will tolerate an initial dose of an mRNA COVID-19 vaccine. We also hypothesize that those individuals experiencing an adverse reaction will tolerate an initial or additional dose of a primary mRNA COVID-19 bivalent vaccine, as indicated.

The study hypothesizes that individuals that have had adverse reactions to a dose of an mRNA COVID-19 vaccine will tolerate an additional dose and those with a personal history of allergic reaction will tolerate vaccination with an mRNA COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria

1. Age over 18.
2. Participant must be able to understand and provide informed consent
3. No evidence of infectious illness (defined as fever >38⁰C, vomiting, diarrhea, new cough, new shortness of breath, new congestion, new runny nose, new headache or sore throat) within 14 days of vaccine administration.
4. Subjects must have a history of adverse reaction to either the Pfizer-BioNTech mRNA COVID vaccination or the Moderna mRNA COVID vaccination, a personal history of allergic reaction without prior mRNA COVID vaccination, or a history of adverse reaction to natural COVID infection.
5. Females of childbearing potential must have a negative pregnancy test prior to vaccination.

Exclusion Criteria

1. Under age 18
2. Inability or unwillingness of a participant to give written informed consent
3. Evidence of COVID-19 infection within 21 days of vaccination visit
4. History of antibody agent or convalescent plasma for treatment or prevention of COVID-19 within 90 days
5. Individuals with known history of a severe allergic reaction (e.g., anaphylaxis) to any component of the Pfizer-BioNTech mRNA COVID-19 vaccination or the Moderna mRNA COVID-19 vaccination.
6. History of underlying immune disorder.

   * Pregnancy
   * Immunocompromised

     * Persons with primary or acquired immunodeficiency
     * Persons on anti-rejection therapy following solid organ transplant or bone marrow transplant
     * Persons on biologic therapeutic agents
     * Persons with malignancy and ongoing or recent chemotherapy
     * Persons receiving systemic immunosuppressive therapy, including corticosteroids equivalent to 20 mg/day of prednisone for 2 weeks
   * Persons with chronic kidney disease stage 3 or higher
   * Persons with history of significant pulmonary compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Percent of participants that have a reaction to an initial or additional dose of the Pfizer-BioNTech or Moderna COVID-19 mRNA vaccine | up to approximately 7 days after the vaccine is given
Number of participants with treatment-related allergic reaction adverse events | up to approximately 7 days after the vaccine is given
  The safety of administering an initial or additional dose will be determined by using the grading of systemic allergic reactions will be based on a scale of 1-5 according to criteria set forth in the Consortium of Food Allergy Research (CoFAR) grading scale (version 3.0) modified for adults as well as the Brighton Collaboration to grade the diagnostic certainty of anaphylaxis.

SECONDARY OUTCOMES:
Number of clinical adverse reaction types (non-allergic) | up to approximately 7 days after the vaccine is given
  The study will grade the severity of non-allergic adverse events experienced by the study participants according to the criteria set forth in the FDA Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007); hereafter, referred to as the FDA Toxicity Grading Scale. Adverse events will be graded on a scale from 1 to 5 according to the following standards in the FDA Toxicity Grading Scale.

CONTACTS AND LOCATIONS:
Overall Officials: James Baker, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No